CLINICAL TRIAL: NCT04478643
Title: Clinical and Microbiological Efficacy of Lactobacillus Reuteri in the Supportive Therapy of Periodontitis: a 6 Months Randomized Controlled Trial
Brief Title: Lactobacillus Reuteri in the Supportive Therapy of Periodontitis
Acronym: PERIOPRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, Magda Mensi, Principal investigator, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PERIOPRO np.: 3965
Record Dates: First submitted 2020-07-06; First posted 2020-07-21 (Actual); Results first posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-06

CONDITIONS: Periodontal Diseases
Keywords: Lactobacillus reuteri; Probiotic; Periodontal diseases; GBT
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Intervention Model Description: Monocentric, Parallel-Arm, Patient, Statistician, Operator and Examiner are blinded, RCT
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PLACEBO (Placebo Comparator): * Collection of microbiological samples from the two deepest sites in two different quadrants.
  * All patients receive full periodontal charting, full mouth periodontal treatment and OHI (oral hygiene instruction).
  * Study lozenges without live bacteria are administered to consume at home. The patients are instructed to dissolve the lozenges on their tongue twice a day, preferably after brushing, for 3 weeks.
  Interventions: Dietary Supplement: Placebo
- PROBIOTIC (L. Reuteri) (Experimental): * Collection of microbiological samples from the two deepest sites in two different quadrants.
  * All patients receive full periodontal charting, full mouth periodontal treatment and OHI (oral hygiene instruction).
  * Study lozenges containing Lactobacillus Reuteri are administered to consume at home. The patients are instructed to dissolve the lozenges on their tongue twice a day, preferably after brushing, for 3 weeks.
  Interventions: Dietary Supplement: Probiotic: Lactobacillus Reuteri

INTERVENTIONS:
Dietary Supplement: Probiotic: Lactobacillus Reuteri — Lactobacillus reuteri ATCC PTA 5289 (a minimum of 2 × 108 colony-forming units L. reuteri Prodentis/lozenge, BioGaia AB)
  Arms: PROBIOTIC (L. Reuteri)
Dietary Supplement: Placebo — Placebo lozenge. Will be identical in taste, texture and appearance to the Probiotic one.
  Arms: PLACEBO

SUMMARY:
Literature shows the potential effectiveness of L. reuteri as an adjunct to non-surgical periodontal therapy in initial treatment of periodontitis, but also underlines the limits of the conclusions, and the heterogeneity and limited sample size of the available studies. Therefore, there is a need for longer-term, randomized, controlled studies. Moreover, only one study addresses the use of this probiotic during the supportive therapy, in particular in patients with severe forms of periodontitis, and only few patients were included.

Patients meeting the criteria of periodontitis stage III and IV, grade C are considered to be affected by severe and advanced forms of periodontitis with a rapid rate of progression. This group of patients could particularly benefit from supplements for the maintenance of periodontal health.

The hypothesis of the present randomized controlled trial is that the adjunctive use of probiotic treatment can bring clinical and microbiological advantages during the supportive therapy of periodontal disease, and reduce the number of residual pockets.

To test this hypothesis, the patients, upon initial evaluation, will be divided in 2 study groups and, after a session of professional oral hygiene, will be prescribed one of the therapies below:

* PLACEBO: The patients of the control group will receive control lozenges without live bacteria;
* TEST: The patients of the probiotic group will receive probiotic lozenges containing Lactobacillus reuteri DSM 17938 and Lactobacillus reuteri ATCC PTA 5289 (a minimum of 2 × 108 colony-forming units L. reuteri Prodentis/lozenge, BioGaia AB).

The probiotic and control lozenges will be identical in taste, texture and appearance. The lozenges will be given to all patients to consume at home. The patients will be instructed to dissolve them on their tongue twice a day, preferably after brushing, for 3 weeks.

Periodontal and microbiological parameters will be evaluated at 3 and 6 months after the initial therapy, and compared between the two groups.

DETAILED DESCRIPTION:
Probiotics are defined as 'live microorganisms which, when administered in adequate amounts, confer a health benefit on the host'. The influence of probiotics on pathogens flora can derive from three principal modes of action: innate and acquired host defense modulation, production of antibacterial substances and competitive exclusion mechanism. In particular, Lactobacillus reuteri has been studied for its antibacterial and anti-inflammatory properties.

It is a heterofermentative bacterium and the distinct strains have different characteristics. In particular it acts as an antibiotic, induces oxidative stress on pathogens, is resistant to proteolytic and lipolytic and present anti-inflammatory properties.

TRIAL DESIGN Parallel-arm, mono-center, statistician operator and examiner blinded RCT. The trial will have 6 months of duration.

STUDY POPULATION Forty-four (44) adults, aged 18-75 years, meeting the criteria of periodontitis stage III and IV, grade C, will be entered into study. It is expected that forty (40) subjects will complete the study.

PRIMARY OUTCOMES

- Change in (Pocket Probing Depth) PPD: change in mean value for each patient will be calculated. Baseline values will be compared to the values recorded at follow-up visits.

SECONDARY OUTCOMES

* Pocket closure
* Risk of progression of periodontitis
* Change in BoP: change in percentage of sites positive to bleeding on probing.
* Change in Plaque Index (PI): change in percentage of sites with presence of plaque. Baseline values will be compared to the values recorded at follow-up visits.
* Change in Periodontal Attachment Level (PAL): change in mean value for each patient will be calculated. Baseline values will be compared to the values recorded at follow-up visits.
* Change in Recession (REC): change in mean value for each patient will be calculated. Baseline values will be compared to the values recorded at follow-up visits.
* Changes in microbial composition and proportion of sequences identified as Lactobacillus reuteri in the deepest residual pockets

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form.
* Male and female subjects, aged 18-75 years, inclusive.
* Good general health (free of systemic diseases such as diabetes, HIV infection or genetic disorder, ongoing malignant disease of any type that could influence the outcome of the treatment and might interfere with the evaluation of the study objectives).
* History of periodontitis staging III or IV grading B or C
* At least 2 sites with probing depth ≥6 mm or pockets of 5 mm with bleeding on probing in two different quadrants.
* Previous periodontal non-surgical treatment at least 3 months maximum 6 months.
* Availability for the 6-month duration of the study for an assigned subject.

Exclusion Criteria:

* Not willing to follow the agreed protocol.
* Presence of orthodontic appliances.
* Smokers (more than 10 cigarettes per day)
* Chronic obstructive pulmonary disease and asthma.
* Tumors or significant pathology of the soft or hard tissues of the oral cavity.
* Current radiotherapy or chemotherapy.
* Pregnant or lactating women.
* Current or past (within 3 months prior to enrolment) administration of medications that may influence periodontal conditions and/or interfere with healing following periodontal treatment (i.e., corticosteroids, calcium channel blockers, systemic antibiotics, ...).
* History of allergy to Erythritol or chlorexidine.
* Restorations on the teeth to be treated which may interfere with treatment administration and/or scoring procedures, at the discretion of the examiner.
* Use of systemically administered antibacterial agents or probiotics 3 months prior to enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2024-02-12 (Actual); Study Completion 2024-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Magda Mensi, Principal Investigator — ASST Spedali Civili di Brescia
Locations (1):
- Magda Mensi, Brescia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- PLACEBO: * Collection of microbiological samples from the two deepest sites in two different quadrants.
  * All patients receive full periodontal charting, full mouth periodontal treatment and OHI (oral hygiene instruction).
  * Study lozenges without live bacteria are administered to consume at home. The patients are instructed to dissolve the lozenges on their tongue twice a day, preferably after brushing, for 3 weeks.
  Placebo: Placebo lozenge. Will be identical in taste, texture and appearance to the Probiotic one.
- PROBIOTIC (L. Reuteri): * Collection of microbiological samples from the two deepest sites in two different quadrants.
  * All patients receive full periodontal charting, full mouth periodontal treatment and OHI (oral hygiene instruction).
  * Study lozenges containing Lactobacillus Reuteri are administered to consume at home. The patients are instructed to dissolve the lozenges on their tongue twice a day, preferably after brushing, for 3 weeks.
  Probiotic: Lactobacillus Reuteri: Lactobacillus reuteri ATCC PTA 5289 (a minimum of 2 × 108 colony-forming units L. reuteri Prodentis/lozenge, BioGaia AB)
Period: Overall Study
Arm/Group | PLACEBO | PROBIOTIC (L. Reuteri)
Started | 22 | 22
Completed | 20 | 20
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PLACEBO | PROBIOTIC (L. Reuteri) | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 20 | 37
  >=65 years | 3 | 0 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.418 (7.765) | 51.961 (12.627) | 51.689 (10.343)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 8 | 8 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 20 | 38
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 18 | 20 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in PD (Periodontal Depth)
Description: Change in mean PD value for each patient measured (from the gingival margin to the bottom of the pocket). Baseline values will be compared to the values recorded in the follow-up visits.
Time Frame: baseline, 3 and 6 months
Measure: Mean (95% Confidence Interval); unit: millimeter
Arm/Group | PLACEBO | PROBIOTIC (L. Reuteri)
Number analyzed (Participants) | 20 | 20
millimeter
  BASELINE | 5.63 [5.24 to 6.05] | 5.45 [5.06 to 5.86]
  3 MONTHS | 4.01 [3.73 to 4.32] | 4.03 [3.75 to 4.33]
  6 MONTHS | 3.92 [3.65 to 4.22] | 3.97 [3.69 to 4.27]

2. Secondary Outcome: Risk Progression of the Periodontitis and the Need of Periodontal Surgery
Description: Change in percentage of patient who need periodontal surgery. Periodontal stability is defined as < 10% of sites bleeding on probing, no probing depths of 4 mm or greater that bleed on probing, and lack of progressive periodontal destruction. Baseline values will be compared to the values recorded in the follow-up visits.
Time Frame: 6 months
Reporting Status: Not Posted

3. Secondary Outcome: Pocket Closure
Description: Change in percentage of site > 4mm. Baseline values will be compared to the values recorded in the follow-up visits.
Time Frame: baseline, 3 and 6 months
Measure: Mean (95% Confidence Interval); unit: percentage
Arm/Group | PLACEBO | PROBIOTIC (L. Reuteri)
Number analyzed (Participants) | 20 | 20
percentage
  BASELINE | 10.7 [7.0 to 16.6] | 9.6 [6.2 to 14.8]
  3 MONTHS | 4.8 [3.0 to 7.5] | 5.9 [3.8 to 9.2]
  6 MONTHS | 5.2 [3.3 to 8.1] | 5.5 [3.6 to 8.7]

4. Secondary Outcome: Microbiological Changes
Description: changes in microbial composition (kind of bacteria) and proportion (% of pathogen) of sequences identified as Lactobacillus reuteri in the deepest residual pockets
Time Frame: baseline, 3 and 6 months
Reporting Status: Not Posted

5. Secondary Outcome: Change in REC (Clinical Gingival Recession)
Description: Change in mean of REC value for each patient should be calculated. Baseline values will be compared to the values recorded in the follow-up visits.
Time Frame: baseline, 3 and 6 months
Measure: Mean (95% Confidence Interval); unit: millimeter
Arm/Group | PLACEBO | PROBIOTIC (L. Reuteri)
Number analyzed (Participants) | 20 | 20
millimeter
  BASELINE | 0.45 [0.18 to 1.12] | 0.51 [0.21 to 1.27]
  3 MONTHS | 0.62 [0.25 to 1.55] | 0.54 [0.22 to 1.34]
  6 MONTHS | 0.76 [0.31 to 1.91] | 0.48 [0.20 to 1.20]

6. Secondary Outcome: Change in CAL (Clinical Attachment Level)
Description: Change in mean of CAL value for each patient should be calculated. Baseline values will be compared to the values recorded in the follow-up visits.
Time Frame: baseline, 3 and 6 months
Measure: Mean (95% Confidence Interval); unit: millimeter
Arm/Group | PLACEBO | PROBIOTIC (L. Reuteri)
Number analyzed (Participants) | 20 | 20
millimeter
  BASELINE | 5.92 [5.45 to 6.44] | 5.79 [5.32 to 6.31]
  3 MONTHS | 4.28 [3.93 to 4.66] | 4.41 [4.05 to 4.80]
  6 MONTHS | 4.17 [3.83 to 4.54] | 4.41 [4.05 to 4.80]

7. Secondary Outcome: Change in BOP (Bleeding on Probing)
Description: Change in percentage of sites positive to bleeding on probing. Baseline values will be compared to the values recorded in the follow-up visits.
Time Frame: baseline, 3 and 6 months
Measure: Mean (95% Confidence Interval); unit: percentage
Arm/Group | PLACEBO | PROBIOTIC (L. Reuteri)
Number analyzed (Participants) | 20 | 20
percentage
  BASELINE | 89.0 [83.3 to 93.0] | 83.5 [76.2 to 88.9]
  3 MONTHS | 50.9 [40.3 to 61.3] | 49.7 [39.5 to 60.0]
  6 MONTHS | 38.8 [29.2 to 49.3] | 42.3 [32.6 to 52.8]

8. Secondary Outcome: Change in PI (Plaque Index)
Description: Change in percentage of site with plaque. Baseline values will be compared to the values recorded in the follow-up visits.
Time Frame: baseline, 3 and 6 months
Measure: Mean (95% Confidence Interval); unit: percentage
Arm/Group | PLACEBO | PROBIOTIC (L. Reuteri)
Number analyzed (Participants) | 20 | 20
percentage
  BASELINE | 52.1 [40.2 to 63.9] | 38.6 [25.5 to 51.7]
  3 MONTHS | 32.4 [18.6 to 46.3] | 31.4 [19.3 to 43.6]
  6 MONTHS | 26.8 [14.0 to 39.6] | 33.6 [21.3 to 45.9]

ADVERSE EVENTS:
Time Frame: 6 months for each subject
Arm/Group | PLACEBO | PROBIOTIC (L. Reuteri)
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-13): https://cdn.clinicaltrials.gov/large-docs/43/NCT04478643/Prot_SAP_000.pdf